CLINICAL TRIAL: NCT02415361
Title: Follow Ups of Parents With Infants With Cleft Lip and Palate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kim Alexander Tønseth, Head of Department of Plastic and Reconstructive Surgery, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014/17828
Record Dates: First submitted 2015-02-27; First posted 2015-04-14 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Cleft Lip; Cleft Palate
Keywords: Parents; Follow-Up Studies
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (No Intervention): Standard care consists of:
  * a phone call from a CLP-nurse after the referral from the local birth hospital has been received
  * telephone service at parents request and at the staffs availability
  * invitation to a one-day-information course before surgery
- Arm B (Active Comparator): Systematic follow up by a special trained nurse consists of:
  * telephone contact with the parents shortly after birth
  * visit at the maternity ward within 36 hours after the referral has been received
  * telephone follow ups at specific times and at parents request
  * guidance and support in feeding and treatment
  * written information
  * cooperation with the staff at the maternity unit and the health centre
  * follow up in accordance with a check-list and log
  * invitation to a one-day-information course before surgery
  Interventions: Other: Cleft lip and palate

INTERVENTIONS:
Other: Cleft lip and palate — Comparison between Arm A who will receive standard care and Arm B who will receive systematic follow up performed by a special trained nurse will be performed.
  Arms: Arm B

SUMMARY:
In Norway, 100-120 children are born with CLP (1.9 per 1,000 live births) each year. Parents of infants with CLP need information and support, especially with feeding immediately after birth. These needs are often not met. The purpose of this study is to investigate the effect of systematic follow ups of parents with infants with CLP performed by a special trained nurse. Parental information needs, parental coping and stress and infant growth and feeding will be explored and compared to a control group receiving standard care. 26 parents (mothers and fathers) or more shall be included in each group according to specific criteria. The control should be examined first. Both groups will answer questionnaires 3 times during the child's first year.

ELIGIBILITY:
Inclusion Criteria:

* Parents of infants with cleft lip and palate (CLP); cleft lip, cleft palate or cleft lip and palate
* Birthplace in south-east region of Norway
* Scandinavian speaking parents

Exclusion Criteria:

* Parents of infants with CLP who are referred to the hospital after the first measure point
* Birthplace outside south-east region of Norway
* Non-scandinavian speaking parents

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Parental stress as measured by Parenting Stress Index (PSI), Perceived Stress Scale (PSS) | 1 month post partum
  Both groups
Parental coping as measured by Post-Discharge Coping Difficulty Scale (PDCDS) | 1 month post partum
  Both Groups
Quality of discharge teaching as measured by Quality of Discharge Teaching Scale (QDTS)-Parent form | 1 month post partum
  Both groups
Infant growth as measured by "Demographic data Questionnaire" and "Child health card" | 1 month post partum
  Both groups
Infant feeding as measured by Survey of infant diets and "Feeding Questionnaire" (study specific questionnaire) | 1 month post partum
  Both groups
Parental stress as measured by Parenting Stress Index (PSI), Perceived Stress Scale (PSS) | 6 months post partum
  Both groups
Infant feeding as measured by Survey of infant diets and "Feeding Questionnaire" (study specific questionnaire) | 6 months post partum
  Both groups
Parental stress as measured by Parenting Stress Index (PSI), Perceived Stress Scale (PSS) | 13 months post partum
  Both groups
Infant growth as measured by "Child health card" | 13 months post partum
  Both groups
Infant feeding as measured by Survey of infant diets and "Feeding Questionnaire" (study specific questionnaire) | 13 months post partum
  Both groups
Parental views on the follow up as measured by "Response on the follow up" (study specific questionaire) | 6 months post partum
  Both groups

CONTACTS AND LOCATIONS:
Overall Officials: Kim A Tønseth, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo university hospital; Rikshospitalet, Oslo, Norway